CLINICAL TRIAL: NCT06171854
Title: A Phase II Trial Evaluating the Activity of caBozantinib in Pre-treated pAtients With Metastatic COlorectal Cancer (mCRC). ABACO Trial.
Brief Title: caBozantinib in Pre-treated pAtients With Metastatic COlorectal Cancer.
Acronym: ABACO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Fortunato Ciardiello, Professor, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMP-001
Record Dates: First submitted 2023-10-26; First posted 2023-12-15 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Refractory Colorectal Adenocarcinoma
Keywords: crc
MeSH Terms: conditions — Colonic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cabozantinib (Experimental): 60 mg once daily. Route: per os Cycle: 28 days
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — cabozantinib in patients with refractory mCRC
  Other Names: Cabometyx

SUMMARY:
This is a phase II non-randomised and non-comparative study, in pretreated mCRC patients, progressed after at least 2 lines of prior chemotherapy for metastatic disease.

Treatment plan:

* First Stage: A total of 22 patients will be enrolled in the first stage to detect at least 3 patients free of progression at 16 weeks
* Second Stage: If at least 3 patients will be free of progression at 16 weeks, an additional cohort of 11 patients will be enrolled in the second stage

DETAILED DESCRIPTION:
The prognosis of patients diagnosed with metastatic colorectal cancer (mCRC) remains poor despite significant progress made in the treatment efficacy and tolerability. The introduction of cytotoxic drugs (i.e. oxaliplatin, irinotecan, and trifluridine/tipiracil) and molecular targeted agents (i.e. bevacizumab, cetuximab, panitumumab, aflibercept, and regorafenib), has dramatically improved patients outcomes with an increase in median overall survival from 6 months with best supportive care only, to more than 30 months with new treatment strategies. The recent advances in genomic technologies have provided further insight into the profound complexity and molecular heterogeneity of colorectal cancer. According to the recent Consensus on CRC Molecular Subtypes (CMS) four biologically distinct subtypes have been identified.

CMS1 (14%) occurring more often in older age, female patients, is characterized by right-sided tumors, hypermutated, enriched for MSI and BRAF mutant and with immune pathway activation. CMS2 (37%) shows epithelial phenotype, left-sided location, chromosomal instability (CIN), microsatellites stable (MSS), TP53 mutation, WNT/MYC pathway activation, and Epidermal Growth Factor Receptor (EGFR) upregulation and is associated with better survival rates; CMS3(13%), also expressing epithelial phenotype, is highly heterogeneous in CIN/MSI status and KRAS and PIK3CA mutant; CMS4 (23%) is defined by mesenchymal phenotype, increased TGF-β and AXL signalling, younger age at diagnosis, invasive phenotype, NOTCH3/VEGFR2 overexpression, and worse survival outcomes. This knowledge cannot be immediately translated into clinical practice, since CMS is not yet used to stratify patients for anti-cancer treatment. However, a better understanding of the complex molecular landscape in CRC will contribute to new treatment strategies.

Cabozantinib is an oral, small-molecule inhibitor of tyrosine kinases, including MET, VEGF receptor 2 (VEGFR2), AXL and RET, currently approved for the treatment of patients with progressive, metastatic medullary thyroid cancer; treatment-naïve patients with renal cell carcinoma with intermediate or poor risk disease or previously treated with a vascular endothelial growth factor (VEGF)-inhibitor; hepatocellular carcinoma (HCC) previously treated with sorafenib.

Angiogenesis is a crucial mechanism in CRC development and progression Moreover, AXL and MET signalling pathways are implicated in CRC invasion and metastasis and are involved in drug resistance occurrence .

Cabozantinib has shown antitumor activity in preclinical CRC patient-derived tumor xenograft (PDTX) model leading to a decrease in the phosphorylation of Tie2, VEGFR2 (pro-angiogenic factors) and the MET, RET and AXL receptors (oncogenic pathways).

ELIGIBILITY:
Inclusion Criteria:

Histologically proven diagnosis of colorectal adenocarcinoma. 2. Male or female patients ≥ 18 years of age. 3. Diagnosis of metastatic disease. 4. Known RAS status (NRAS and KRAS exon 2,3 and 4) per local laboratory assessment.

5. Patients should have received at least two standard lines of treatment including all the following: fluoropyrimidines, irinotecan, oxaliplatin, anti-angiogenic drugs (eg. bevacizumab and or aflibercept) and, in case of patients harbouring RAS WT tumours, anti-Epidermal Growth Factor receptors monoclonal antibodies (cetuximab or panitumumab). Note: Prior treatment with trifluridine-tipiracil is allowed.

6. Recovery to baseline or ≤ Grade 1 CTCAE v.5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.

7. Measurable disease according to RECIST criteria v1.1. 8. ECOG Performance Status 0-1. 9. Life expectancy of at least 3 months. 10. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 10 days before study entry:

* Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L).
* Platelets ≥ 100,000/mm3 (≥ 100 GI/L).
* Hemoglobin ≥ 9 g/dL.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 × upper limit of normal.
* Total bilirubin ≤ 1.5 × the upper limit of normal. For subjects with Gilbert's disease ≤ 3 mg/dL.
* Fasting serum triglycerides ≤ 2.5 × upper limit of normal and total cholesterol ≤ 300 mg/dL.

Note: Lipid-lowering medication is allowed.

* HbA1c ≤ 8%.
* Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockroft-Gault equation.
* 24-hour urine protein < 1 g. 11. In the investigator judgement, compliance with the protocol requirements and signed informed consent document. 12. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.

  13. Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, low body weight, ovarian suppression or other reasons.

Exclusion Criteria:

Prior treatment with cabozantinib. 2. Prior treatment with VEGFR-targeting TKI (e.g. regorafenib). 3. Treatment with any anticancer drug within 4 weeks before study entry. 4. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before study entry. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.

5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before study entry. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of study entry.

6. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel).

Note: Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (<1 mg/day), and low dose, low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 12 weeks before study entry, and who have had no complications from a thromboembolic event or the anticoagulation regimen.

7. Chronic treatment with corticosteroids or other immunosuppressive agents (with the exception of inhaled or topical corticosteroids or corticosteroids with a daily dosage equivalent ≤ 10 mg prednisone). Subjects with brain metastases requiring systemic corticosteroid are not eligible.

8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

* Cardiovascular disorders:

  * Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
  * Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
  * Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before study entry.
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
  * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before study entry. Note: Complete healing of an intra-abdominal abscess must be confirmed before study entry.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of redblood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before study entry.
* Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.
* Lesions invading major pulmonary blood vessels.
* Other clinically significant disorders such as:

  * Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)- related illness, or chronic hepatitis B or C infection.
  * Serious non-healing wound/ulcer/bone fracture.
  * Malabsorption syndrome.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ transplantation. 9. Major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 3 months before study entry. Complete wound healing from major surgery must have occurred 1 month before study entry and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before study entry. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.

    10. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec within 1 month before study entry.

    11. Pregnant or lactating females. 12. Inability to swallow tablets. 13.Previously identified allergy or hypersensitivity to components of the study treatment formulation.

    14. Diagnosis of another malignancy within 2 years before study entry, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 16 weeks
  Progression Free Survival (PFS) rate at 16 weeks: the rate of patients who have not experienced disease progression or death for any cause at 16 weeks.

SECONDARY OUTCOMES:
Progression Free survival (PFS) | from the start of the study treatment until disease progression or death for any cause, assessed up to 100 months
  calculated from the start of the study treatment until disease progression or death for any cause.
Overall Survival (OS) | from the start of the study treatment until death for any cause, assessed up to 100 months
  calculated from the start of the study treatment until death for any cause.
Response Rate | rate of patients with complete response or partial response, as best response, through study completion, an average of 1 year
  rate of patients with complete response or partial response, as best response.
Disease Control Rate (DCR) | rate of patients with complete response, partial response and stable disease, as best response, during the course of the study, average time one year
  rate of patients with complete response, partial response and stable disease, as best response.
Safety as the description of adverse events | through study completion, an average of 1 year
  Adverse events graded according Criteria for Adverse Events (CTCAE) Version(v.) 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Martinelli, MD, PhD, Principal Investigator — erika.martinelli@unicampania.it
Locations (1):
- A.O.U dell'Università degli Studi della Campania "Luigi Vanvitelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No